CLINICAL TRIAL: NCT00000250
Title: Cold Water Immersion Modulates Reinforcing Effects of Nitrous Oxide
Brief Title: Cold Water Immersion Modulates Reinforcing Effects of Nitrous Oxide - 2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: NIDA-08391-2; R01DA008391 (NIH); R01-08391-2
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Opioid-Related Disorders; Substance-Related Disorders
Keywords: nitrous oxide; choice; subjective effects; pain; analgesia; reinforcer; healthy volunteer
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders; Pain; Agnosia

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Lukewarm water (Active Comparator): Subjects will immerse forearm in lukewarm water while inhaling 0% and 40% N2O in 2 sampling trials, then choose between intervntions for one choice trial
  Interventions: Drug: 0% N2O; Drug: 40% N2O
- Ice cold water (Active Comparator): Subjects will immerse forearm in ice cold water while inhaling 0% and 40% N2O in 2 sampling trials, then choose between intervntions for one choice trial
  Interventions: Drug: 0% N2O; Drug: 40% N2O

INTERVENTIONS:
Drug: 0% N2O — Subjects will inhale 100% oxygen with no N2O for 25 min then immerse forearm in warm water and cold water
Drug: 40% N2O — Subjects will inhale 40% N2O then immerse forearm in warm water and cold water

SUMMARY:
The purpose of this study is to conduct experiments to examine subjective and reinforcing effects of nitrous oxide. Mood altering and psychomotor effects will be tested on non-drug abusers and preference procedures will be used to assess reinforcing effects. To evaluate: cold water immersion modulates the reinforcing effects of nitrous oxide in healthy volunteers.

ELIGIBILITY:
Please contact site for information.

Ages: 21 Years to 32 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 1993-12; Primary Completion 1995-05 (Actual); Study Completion 1995-05 (Actual)

PRIMARY OUTCOMES:
Subject's choice of intervention | After sampling trials

CONTACTS AND LOCATIONS:
Overall Officials: James Zacny, Ph.D., Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Anesthesia & Critical Care, Chicago, Illinois, United States

REFERENCES:
- [Background] Experimentall Clinical Psycopharmacoly 1995, 3(2):148-155